CLINICAL TRIAL: NCT01735812
Title: Cryoablation of Symptomatic Uterine Fibroids Using the IceSense3™ System in a Percutaneous Laparoscopic-assisted Approach
Brief Title: Laparoscopic Cryoablation of Uterine Fibroids
Acronym: UFREEZE-01
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: IceCure Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICUFL-01
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2012-11

CONDITIONS: Symptomatic Uterine Fibroids
Keywords: cryoablation; uterine fibroid; uterine myoma; who completed her family planning; but wishes to preserve her uterus
MeSH Terms: conditions — Leiomyoma; Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- symptomatic UF (Experimental)
  Interventions: Device: IceSense3 system

INTERVENTIONS:
Device: IceSense3 system — The IceSense3™ is a modern cryosurgical device that was designed by IceCure Medical for a variety of applications.

SUMMARY:
The goal of this study is to evaluate the safety & efficacy of cryoablation using IceCure medical's IceSense3™ device for the treatment of symptomatic uterine fibroids in a percutaneous lap-assisted approach.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal woman between the ages of 30 and 50 (inclusive)
2. Patient had completed her family planning and does not desire future childbearing.
3. Patient is suffering from menorrhagia as a result of symptomatic uterine fibroids.
4. Patient's uterus size is smaller than 18 gestational weeks.
5. Patient wishes to preserve her uterus and avoid hysterectomy.
6. Patient has 1-3 treatable uterine fibroids in size of up to 10cm measured by US/MRI.
7. Overall treated fibroid volume is ≤ 3,138cm3 (width x length x height x 0.523)
8. Patient has clinical menorrhagia as indicated by menstrual blood loss of ≥160 ml during one baseline cycle prior to treatment.
9. Patient is able to visit the clinic as needed during the 1 year follow-up period following the treatment.
10. The patient has been informed of the study and agrees to its provisions, and has signed an IRB approved written informed consent, including data privacy authorization.

Exclusion Criteria:

1. Patient had not finished her family planning
2. Patient was already treated for uterine fibroids in the past (UAE, myomectomy, HIFU,…) or undergone endometrial ablation.
3. Patient had been treated with GnRH over the last 3 months.
4. Patient has known symptomatic endometriosis that cannot be completely removed during laparoscopic procedure.
5. Patient has known or suspected adenomyosis
6. Patient had any active abdominal/pelvic inflammatory disease.
7. Patient has known or suspected gynecologic malignancy.
8. Patient with submucosal fibroids type "zero"
9. Patient with undiagnosed vaginal bleeding
10. Patient with blood clotting disorders
11. Patients carrying contagious diseases such as Tuberculosis Hepatitis or AIDS.
12. Patient participating in other trials using drugs or devices.
13. Patient is unable to commit all study requirements including follow-up visits and questionnaires.
14. Patient has any contraindication for laparoscopic surgery

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement in patient's fibroid-related quality of life | 12 months
  To evaluate procedural efficacy by the improvement in patient's fibroid-related quality of life as assessed in scores of symptom severity subscale questionnaire (SSS-UFS-QOL) at 12 months post-treatment comparing to baseline score.
Incidence, subsequent interventions and procedure-related adverse events | 12 months
  To evaluate procedural safety by monitoring incidence, subsequent interventions and procedure-related adverse events within 12 months of treatment

SECONDARY OUTCOMES:
Reduction in fibroid volume | 12 months
  Reduction in fibroid volume as measured by US/MRI imaging at 6 and 12 months follow-up post treatment comparing to baseline.
Improvement in menstrual bleeding | 12 months
  Improvement in menstrual bleeding compared to baseline as measured in chemical analysis (Alkaline haematin technique) at 6 and 12 months post treatment.
Improvement in patient's fibroid-related quality of life | 6 months
  Improvement in patient's fibroid-related quality of life as assessed in scores of symptom severity subscale questionnaire (SSS-UFS-QOL) at 6 months post-treatment comparing to baseline score.

OTHER OUTCOMES:
Patient's and physician's overall treatment evaluation | 12 months
  Patient's and physician's overall treatment evaluation and satisfaction will be assessed using a self-report questionnaire at 6 and 12 months post treatment.
Patient blood loss | 12 months
  Patient blood loss will be also evaluated by Hemoglobin (Hb) level measurements at 6 and 12 months post treatment and will be compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Moty Pansky, Prof., Principal Investigator — Assaf Harofe Hospital, Israel
Locations (1):
- Assaf Harofe, Zrifin, Israel